CLINICAL TRIAL: NCT04099862
Title: Eus-giuded Biliary Drainage With Ec-lams vs ERCP as a Primary Intervention for Endoscopic Treatment of Patinets With Distal Malignant Biliary Obstruction
Acronym: EUS-BD
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 2339
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: DISTAL MALIGNANT BILIARY OBSTRUCTION
MeSH Terms: interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ERCP: Endoscopic retrograde cholangiopancreatography (ERCP)
  Interventions: Procedure: ERCP
- EUS-BD: Endoscopic UltraSound Biliary Drainage
  Interventions: Procedure: EUS-BD

INTERVENTIONS:
Procedure: ERCP — Endoscopic retrograde cholangiopancreatography (ERCP)
  Groups: ERCP
Procedure: EUS-BD — Endoscopic UltraSound Biliary Drainage
  Groups: EUS-BD

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) is the gold standard for the management of jaundice in patients with distal malignant biliary obstruction. However, surgically altered anatomy (i.e., Whipple intervention, Roux-en-Y gastric bypass, Billroth II surgery), periampullary diverticula, gastric outlet obstruction, and malignant obstruction of the lumen determine the failure of the procedure in about 5-10% of cases, requiring alternative methods of decompression. Percutaneous transhepatic biliary drainage (PTBD) and surgical bypass are well established alternatives in these patients, but associated with increased morbidity, longer length of hospital stay and higher costs.

EUS guided biliary drainage (EUS-BD) through a transduodenal access is an alternative in cases of failed or unfeasible ERCP. EUS-BD has considerably evolved thanks to the development of dedicated devices such as lumen apposing metal stents (LAMS), specifically designed for endoscopic ultrasound procedures. LAMS are made up of braided nitinol that is fully covered with silicone to prevent tissue ingrowth, with wide flanges on both ends to provide anchorage.

Recently, LAMS have been incorporated into a delivery system with an electrocautery mounted on the tip (Hot Axios; Boston Scientific Corp.), which allows the device to be used directly to penetrate the target structure without the need to utilize a 19G needle, a guidewire, and a cystotome for prior dilation. This has been described for drainage of peri-pancreatic fluid collections, common bile duct (CBD), gallbladder, and for creation of gastro-jejuno anastomosis. The biliary drainage procedure performed with the Hot Axios sistem is a fast, one-step procedure that obviates the need accessory exchange and thus potentially reduces the risk of complications.

The procedure has been described as safe and effective with a technical success of 98.2%, clinical success of 96.4%, and low rate of complications 7% (consisting of duodenal perforations, bleeding and transient cholangitis).

Patients with distal malignant biliary obstruction have a higher risk of ERCP failure, related to the difficulty of bile duct cannulation or access to the second duodenal portion due to the presence of a stenosis. This condition could imply the need of more advanced cannulation techniques (such as pre-cut, Double Guide Wire DGW technique, pancreatic septotomy) with consequent higher risk of developing post ERCP pancreatitis (PEP). Unlike ERCP, an reaching the papilla is not a requisite for a successful EUS-BD. Moreover, since the papilla is not cannulated and the pancreatic duct is not accessed, this is expected to result in a minimal risk of post-procedural pancreatitis (about 0.50%).

The investigators hypothesize that, in patients with distal malignant biliary obstruction, EUS guided biliary drainage as first step approach has a lower risk of post-procedural pancreatitis compared to standard ERCP. The investoigators propose to perform a randomized controlled study to test this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years

  * Patients with distal malignant biliary obstruction
  * Abdominal ultrasound or computed tomography or magnetic resonance or EUS showing a dilated common bile duct > 15 mm diameter.
  * Agree to receive follow up phone calls
  * Able to provide written informed consent

Exclusion Criteria:

* Coagulation and/or platelets hereditary disorders and/or INR>1.5, PLT<50,000.
* Use of anticoagulants that cannot be discontinued
* Pregnant women
* Inability to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with distal malignant biliary obstruction, who need endoscopic biliary drainage, will be randomized with a 1:1 ratio to undergo jaundice treatment by ERCP or EUS guided biliary drainage.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2021-02-28 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Rate of post-procedural acute pancreatitis | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Endoscopy Unit, Humanitas Research Hospital, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Anderloni A, Spadaccini M, Binda C, Mauro A, Stigliano S, Carrozza L, Colombo M, Mazza S, Coluccio C, Amato A, Andreozzi M, Maria Rizzo GE, Facciorusso A, Radaelli F, Carrara S, Mangiavillano B, Di Matteo FM, Tarantino I, Hassan C, Repici A, Fugazza A, Fabbri C. Endoscopic Ultrasound-Guided Choledochoduodenostomy vs Endoscopic Retrograde Cholangiopancreatography in Malignant Distal Biliary Obstruction to Prevent Postprocedural Pancreatitis: A Randomized Trial. Gastroenterology. 2026 Jan 9:S0016-5085(25)05982-7. doi: 10.1053/j.gastro.2025.09.003. Online ahead of print. PMID 41511419